CLINICAL TRIAL: NCT01101581
Title: Phase I/II Study of Veltuzumab Combined With 90Y-Epratuzumab Tetraxetan in Patients With Relapsed/Refractory, Aggressive Non- Hodgkin's Lymphoma
Brief Title: Study of Veltuzumab and 90Y-Epratuzumab in Relapsed/Refractory, Aggressive NHL
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hA20/90Y-hLL2-01
Record Dates: First submitted 2010-03-16; First posted 2010-04-12 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2020-12

CONDITIONS: Non Hodgkin's Lymphoma; NHL; Aggressive NHL; Diffuse Large B-cell Lymphoma
Keywords: Diffuse Large cell NHL; Mantle cell NHL; Lymphoblastic lymphoma; Diffuse mixed cell lymphoma; Diffuse large cell lymphoma; large noncleaved cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — veltuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Veltuzumab and 90Y-Epratuzumab Tetraxetan (Experimental): Veltuzumab and 90Y-Epratuzumab Tetraxetan target different b-cells. Veltuzumab will be administered in all 4 weekly study drug treatments. 90Y-Epratuzumab Tetraxetan will be administered only on days 8 & 15. The dose of veltuzumab remains the same for all patients.
  Interventions: Drug: Veltuzumab and 90Y-Epratuzumab Tetraxetan; Drug: 90Y-epratuzumab tetraxetan; Drug: veltuzumab
- 90Y-epratuzumab tetraxetan (Experimental): 90Y-epratuzumab tetraxetan will be administered 6 mCi/m2 on days 8 and 15.
  Interventions: Drug: 90Y-epratuzumab tetraxetan

INTERVENTIONS:
Drug: Veltuzumab and 90Y-Epratuzumab Tetraxetan — Veltuzumab will be administered subcutaneously in phase 2. 90Y-Epratuzumab tetraxetan will be administered intravenously. Veltuzumab is given once weekly for 4 weeks. 90Y-Epratuzumab is also given at treatment weeks 2 & 3 (days 8 & 15).
  Other Names: veltuzumab; IMMU-106; hA20; humanized CD20; epratuzumab-tetraxetan; 90Y-hLL2; IMMU-102; humanized CD22
  Arms: Veltuzumab and 90Y-Epratuzumab Tetraxetan
Drug: 90Y-epratuzumab tetraxetan
  Other Names: 90Y-hLL2; 90Y-hLL2-DOTA; 90Y-CD22
Drug: veltuzumab — Veltuzumab will be administered subcutaneously on days 1, 8, 15 and 23
  Other Names: hA20; humanized CD20; IMMU-106
  Arms: Veltuzumab and 90Y-Epratuzumab Tetraxetan

SUMMARY:
The goal of this study is to evaluate a new approach to immunotherapy in NHL by combining two antibodies, veltuzumab and epratuzumab. For treatment, epratuzumab has also been attached to a radioactive isotope called 90yttrium (90Y-epratuzumab). Veltuzumab and 90Y-epratuzumab attack different areas on lymphoma cells. Because of this, treatment with the combination may provide more effective treatment in NHL than either veltuzumab or 90Y-epratuzumab given alone.

DETAILED DESCRIPTION:
The treatment portion of this study consists of study drug administrations each week for four weeks in a row (a total of 4 treatment days). Patients will then return at intervals up to 12 weeks for blood samples and for evaluations to see if their disease responded and to monitor any adverse effects related to treatment. Some blood tests may then need to be repeated at least a few times and/or until any abnormal findings at earlier evaluations have resolved. Otherwise, patients will continue to be evaluated every 3 months for two years, then every 6 months up to 5 years or until the disease worsens. Participation in the study will end when NHL disease worsens.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 years old
* Histological diagnosis of CD20+ B-cell NHL, with DLBCL or other aggressive lymphomas by WHO lymphoma criteria including mantle cell lymphoma and transformed follicular lymphoma.
* Failed at least one prior standard treatment regimen for NHL
* If DLBCL, either received, ineligible for or refused high-dose chemotherapy with stem cell transplant
* Measurable NHL disease by CT, with at least one lesion >1.5 cm in one dimension
* Adequate performance status (>70 Karnofsky scale, 0-1 ECOG)* with an estimated life expectancy of at least 6 months
* Laboratory parameters:

  * Adequate hematology (Hemoglobin >/= 10 g/dL, ANC >/= 1.5 ´ 109/L, platelets >/=100 x 109/L) without ongoing transfusional support
  * Adequate renal and liver function (creatinine and bilirubin </= 1.5 x IULN; AST and ALT </= 2.5 x IULN)
* Otherwise, <Grade 1 toxicity at study entry by NCI CTC version 3.0.
* 3 months beyond any prior rituximab or veltuzumab treatment, 12 weeks beyond autologous stem cell transplant and 4 weeks beyond chemotherapy, other experimental treatments, or any radiation therapy to the index lesion(s).
* Screened for hepatitis B (no time limit) and negative by tests included in NCCN guidelines (hepatitis B surface antigen/antibodies, core antigen/antibodies, hepatitis B e-antigen).
* Patients of childbearing potential must be willing to practice birth control during the study until at least 12 weeks after last veltuzumab infusion; women of childbearing potential must have a negative urine or serum pregnancy test to enter the study.
* Ability to provide signed, informed consent

Exclusion Criteria:

* Pregnant or lactating women. Women of childbearing potential are required to have a negative pregnancy test

  * NCI CTC Grade 3 or 4 infusion reaction to prior anti-CD20 antibodies (rituximab, veltuzumab, etc.)
  * A known anti-antibody response to prior antiCD20 antibodies (HACA positive, HAHA positive, etc)
  * Prior radioimmunotherapy, including Zevalin or Bexxar.
  * Prior high-dose chemotherapy with peripheral blood stem cell transplant.
  * Prior therapy with other human or humanized monoclonal antibodies, unless HAHA tested and negative
  * Primary CNS lymphoma, HIV lymphoma or transformed lymphoma, or presence of symptomatic CNS metastases or carcinomatous meningitis.
  * Rituximab or veltuzumab resistant, defined as having progressed during or within 6 months of any prior rituximab or veltuzumab treatment.
  * Bulky disease by CT, defined as any single mass >10 cm in its greatest diameter
  * Bone marrow involvement ≥25%
  * Prior external beam radiation therapy to >30% bone marrow.
  * Pleural effusion with positive cytology for lymphoma
  * Patients known to be HIV positive, hepatitis B positive, or hepatitis C positive
  * Known autoimmune disease or presence of autoimmune phenomena.
  * Evidence of infection or requiring antibiotics within 7 days.
  * Use of systemic corticosteroids within 2 weeks, except low dose regimens (prednisone, <20 mg/day, or equivalent) which may continue if unchanged.
  * Prior malignancies (other than non-melanoma skin cancer or carcinoma in situ of the cervix) unless disease free for 5 years.
  * Prior malignancy with less than a 5-year disease-free interval, excluding nonmelanoma skin cancers and carcinoma in situ of the cervix.
  * Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Safety/dose limiting toxicity | 12 weeks
  Patients are closely monitored during and after all infusions, and then at intervals over a 12-week post-treatment evaluation period. Safety evaluations required in all patients include vital signs, physical examination, CBC, serum chemistries, serum immunoglobulins, urinalysis, peripheral blood B-cell levels (immunophenotyping based on CD19), and HAHA (to be analyzed by Sponsor). Adverse events and abnormal laboratories will be graded for toxicity according to NCI CTC v3.0 criteria.

SECONDARY OUTCOMES:
Efficacy | 12 weeks-5 years
  CT or PET/CT imaging will be used to quantify changes in index lesions identified on baseline imaging, with responses classified according to revised response criteria for NHL (Cheson, 2007).
  Patients with stable disease or objective responses continue limited follow-up evaluations, including CT evaluations, physical examinations and serum laboratories every 3 months for the first year and then every 6 months up to a total of 5 years or until progression of disease.

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (7):
- United States (7):
  - Helen F. Graham Cancer Center, Newark, Delaware
  - MDACC Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Weill Med College of Cornell Univ/NYH, New York, New York
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Morschhauser F, Leonard JP, Fayad L, Coiffier B, Petillon MO, Coleman M, Schuster SJ, Dyer MJ, Horne H, Teoh N, Wegener WA, Goldenberg DM. Humanized anti-CD20 antibody, veltuzumab, in refractory/recurrent non-Hodgkin's lymphoma: phase I/II results. J Clin Oncol. 2009 Jul 10;27(20):3346-53. doi: 10.1200/JCO.2008.19.9117. Epub 2009 May 18. PMID 19451441
- [Background] Goldenberg DM, Morschhauser F, Wegener WA. Veltuzumab (humanized anti-CD20 monoclonal antibody): characterization, current clinical results, and future prospects. Leuk Lymphoma. 2010 May;51(5):747-55. doi: 10.3109/10428191003672123. PMID 20214444
- [Background] Morschhauser F, Kraeber-Bodere F, Wegener WA, Harousseau JL, Petillon MO, Huglo D, Trumper LH, Meller J, Pfreundschuh M, Kirsch CM, Naumann R, Kropp J, Horne H, Teoh N, Le Gouill S, Bodet-Milin C, Chatal JF, Goldenberg DM. High rates of durable responses with anti-CD22 fractionated radioimmunotherapy: results of a multicenter, phase I/II study in non-Hodgkin's lymphoma. J Clin Oncol. 2010 Aug 10;28(23):3709-16. doi: 10.1200/JCO.2009.27.7863. Epub 2010 Jul 12. PMID 20625137